CLINICAL TRIAL: NCT01586611
Title: A Multicentre, Randomized, Open Label, Phase III Study of Gemcitabine Versus FOLFOX in the First Line Setting for Metastatic Pancreatic Cancer Patients Using Human Equilibrative Nucleoside Transporter 1 (hENT1) Biomarker Testing.
Brief Title: A Study to See if hENT1 Testing on Tumour Tissue Can Predict Response to Treatment With Gemcitabine Chemotherapy and if a Different Chemotherapy Called FOLFOX is Better Than Gemcitabine in Metastatic Pancreas Cancer
Acronym: Panc001
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Panc001
Record Dates: First submitted 2012-04-24; First posted 2012-04-27 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (Active Comparator): Cycles to be 4 weeks in length Gemcitabine 1000 mg/m2 IV weekly for 3 weeks then one week off
  Interventions: Drug: Gemcitabine
- FOLFOX (Experimental): Cycles to be 2 weeks in length Oxaliplatin 100 mg/m2 IV day 1 Leucovorin 400 mg/m2 IV day 1 5-FUl 400 mg/m2 IV day 1 5-FU 2400 mg/m2 IV continuous infusion over 46 hours starting day 1
  Interventions: Drug: 5FU, leucovorin, oxaliplatin

INTERVENTIONS:
Drug: 5FU, leucovorin, oxaliplatin — Oxaliplatin 100 mg/m2 IV day 1 Leucovorin 400 mg/m2 IV day 1 5-FUl 400 mg/m2 IV day 1 5-FU 2400 mg/m2 IV continuous infusion over 46 hours starting day 1
  Arms: FOLFOX
Drug: Gemcitabine — 1000 mg/m2 IV weekly for 3 weeks then one week off
  Arms: Gemcitabine

SUMMARY:
Chemotherapy is often used to help shrink the cancer temporarily and may improve survival for patients with incurable pancreas cancer that has spread to other organs. In Canada, the gemcitabine chemotherapy is used to treat pancreas cancer that has spread. The combination of oxaliplatin with other chemotherapies, including 5-fluorouracil, leucovorin, and irinotecan has also been studied and has benefit for patients with advanced pancreas cancer. To date, there is no test that can be done on a patient's tumour to tell if chemotherapy will work in pancreatic cancer. Human equilibrative nucleoside transporter 1 (hENT1) has been shown to be a possible predictor that gemcitabine may or may not work but this needs to be proven in a randomized study where patients get treated with gemcitabine or a different kind of chemotherapy while their tumours get tested for hENT1.

This study is being done because we want to prove that hENT1 can predict if gemcitabine will work in advanced pancreas cancer and if it can, we also would like to show that a different chemotherapy combination called FOLFOX (a combination of 5-fluorouracil, leucovorin, and oxaliplatin) will be helpful for patients whose tumours don't have hENT1.

DETAILED DESCRIPTION:
Pre-clinical and retrospective clinical data indicates hENT1 may be a predictive and prognostic biomarker for gemcitabine (Gem) efficacy. To ultimately prove its use as a biomarker, a prospective randomized study with hENT1 stratification is required. This study would provide the highest level of confidence, and would, if positive, vault Gem into the select few anticancer agents for which a truly sensitive population can be rationally treated. By this "molecular triage", the risk/benefit ratio of Gem therapy for pancreas cancer (PC) could be meaningfully improved while also providing rationale for the use of a different treatment regimen should tumours have low hENT1. The comparator arm of FOLFOX was chosen because of the recent data showing impressive patient outcomes with the use of oxaliplatin-based treatments.

This is a randomized, open-label, multicentre, phase III trial in which eligible patients with metastatic pancreatic adenocarcinoma will be randomized between Gem and FOLFOX with predefined upfront testing for hENT1. To be eligible, patients will have to have adequate tissue available for hENT1 testing which the Cross Cancer Institute (CCI) will ensure prior to treatment randomization. Patients will have their tumour sample tested for the expression of hENT1. A blinded pathologist with expertise knowledge and experience with hENT1 staining at the lead centre (CCI) will be responsible for pathologic hENT1 classification via IHC. hENT1 IHC will be determined and scored as previously outlined.(1) Once hENT1 status has been confirmed, patients will then be randomized 1:1 between Gem and FOLFOX. Patients will be treated on study until disease progression, overwhelming toxicity, or patient withdrawal of consent. Dose adjustments for one or more of the study drugs will be based on toxicities encountered by individual patients. Specific dose-adjustment and treatment guidelines for hematologic and non-hematologic toxicities including neutropenia, diarrhea, renal toxicity, and neurotoxicity will be outlined in the protocol. Prior to enrolment, screening procedures will document compliance with inclusion and exclusion criteria. The primary endpoint will be determination of the difference in PFS in the two study arms, defined from the study start date until either an increase in the sum of the products of the diameters of measurable lesions by ≥ 20% bases on revised RECIST guidelines version 1.1 (2), the appearance of any new lesion, or a deterioration in clinical status that is consistent with disease progression. Secondary endpoints will be determination of the differences in overall response rate (ORR), disease control rate (DCR), and overall survival (OS). Administered dose intensity of Gem and FOLFOX will be reported. Health-related quality of life (HRQL) will be assessed for the duration of active treatment on study.

Patient Population: The target population is patients with measurable metastatic adenocarcinoma of the pancreas who have not been previously treated with systemic therapy for their metastatic disease and who have tumour samples amenable to hENT1 testing. Fine needle aspiration biopsies will not be permitted. Patients who have received prior chemotherapy delivered as part of initial curative therapy (i.e. neoadjuvant, adjuvant, and/or concurrently delivered with radiation and/or surgery) are permitted as long as that treatment was completed at least 6 months prior to study start date. Patients may have received prior radiotherapy or surgery ≥ 4 weeks before study entry and must have recovered from the toxic effects from any prior therapy. Patients with locally advanced adenocarcinoma of the pancreas will be excluded. Full inclusion and exclusion criteria are detailed in the protocol.

Study Objectives:

Primary Objective: To determine the difference PFS between Gem and FOLFOX treated patients in hENT1 high and hENT1 low pancreatic adenocarcinoma.

Secondary Objectives: 1) To determine the difference in ORR between the two treatment arms; 2) To determine the rate of disease control, defined as the sum of complete response rate, partial response rate, and stable disease between the two treatment arms; 3) To determine the difference in OS between the two treatment arms; 4) To determine the differences in HRQL of patients on the two treatment arms.

Exploratory Objectives: 1) To investigate the role of hCNT3 and its interaction with hENT1-related patient outcomes. 2) To evaluate excision repair cross complementing 1 (ERCC1) and microsatellite instability (MSI) in tumour samples, both of which are increasingly being linked to efficacy in oxaliplatin-based therapy but for which information in PC is lacking.

Duration of Treatment: Treatment will continue until objective or symptomatic disease progression, overwhelming toxicity, or patient withdrawal of consent. A patient may continue to receive all or any combination of study drugs for as long as the investigator feels is appropriate, but will be discontinued from study in case of:

1) Clinical and/or radiological documented disease progression (as determined by revised RECIST 1.1 criteria).(2) All drugs will be discontinued and the patient removed from study; 2) Occurrence of unacceptable toxicity (this may be due to one or more drugs resulting in one or more study drug discontinuation); if all three drugs are discontinued the patient will be removed from study; 3) Failure to recover from hematologic and/or non-hematologic toxicity to re-treatment level despite dosing interruption of up to 28 days (this may be due to one or more study drugs resulting in one or more study drug discontinuation); if all drugs in regimen are discontinued the patient will be removed from study; 4) Patient's request (withdrawal of consent) or Investigator's recommendation (this may be one or more study drugs); if all three study drugs are discontinued patient will be removed from study; 5) Patient death (complete Serious Adverse Event Report for deaths occurring within 30 days after last study drug dose OR for deaths occurring after 30 days, only if considered related to study drug).

Efficacy Endpoints: Response assessments will be performed every 8 weeks, regardless of treatment cycle. History, physical exam, laboratory work, imaging, ECOG performance status (PS), will be required at each response assessment. PS will be measured using the ECOG performance status scale. Tumor marker (CA19-9) may be followed at the discretion of the investigator but should not be used in determination of disease response and are not a requirement of the study. Tumor response will be evaluated according to the revised RECIST criteria 1.1.(2) Symptomatic progression will be defined as new or worsening disease symptoms deemed by the treating oncologist to incompatible with continuation of study medication or the requirement for palliative radiation therapy or a fall in ECOG performance status to ≥ 3 deemed to be due to disease and not study treatment. Should symptomatic progression occur, imaging to confirm progression is advised but if not possible due to performance status, the study stop date will be recorded as the date of progression.

Safety: The NCI CTCAE (version 4.0) will be used to evaluate the clinical safety of the treatment in this study. Subjects will be assessed for adverse events at each clinical visit and as necessary throughout the study. Safety will be assessed via vital signs, physical exams, laboratory tests (including hematologic, serum chemistry, and liver function testing), and adverse event determination. Pregnant and nursing females will be excluded from participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic pancreatic adenocarcinoma not previously treated with palliative systemic therapy
* Metastatic disease based on the presence of clinically and/or radiologically documents Measurable disease base on RECIST.
* Adequate tissue (core biopsy) available for IHC testing of hENT1. This may be from primary tumour or metastatic site. Fine needle aspiration biopsies will not be allowed. Histological/cytological confirmation of tissue to ensure sufficient material is available for hENT1 analysis by the Cross Cancer Institute is required prior to starting a patient on study. Biopsies from metastatic sites must be obtained ≥ 3 months after any adjuvant chemotherapy (if applicable). If a patient has had previous surgical resection of their primary tumours, that tissue can be utilized. Tissue sufficient for preparing ≥ 10 unstained slides for central storage and testing is required.
* ECOG performance status of 0 - 1.
* Age ≥ 18 years.
* Life expectancy of at least 3 months based on discretion of treating oncologist.
* Adequate hematologic function defined by the following laboratory parameters:
* Hemoglobin ≥ 100
* Platelet count ≥ 100
* Absolute granulocyte count ≥ 1.5
* Adequate hepatic and renal function defined by the following laboratory parameters:
* AST and ALT ≤ 2.5 X upper limit of institutional normal (≤ 5 if liver metastases)
* bilirubin ≤ upper limit of institutional normal
* calculated creatinine clearance of ≥ 50 mL/min using the Cockcroft-Gault formula, if just below 50 mL/min based on this formula then GFR ≥ 50 mL/min as determined by 24 hr urine collection
* Patients who have received prior chemotherapy or radiation delivered as part of initial curative therapy (i.e. neoadjuvant or adjuvant chemotherapy administered alone and/or concurrently delivered with radiation and/or surgery) are permitted as long as that treatment was completed at least 6 months prior to study start date.
* Patients may have received prior palliative radiotherapy (unless radiation was curative therapy to pelvis or to ≥ 25% of bone marrow stores) if this radiation was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment
* Patients may have received prior surgery if this surgery was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.

Exclusion Criteria:

* Patients who have received prior palliative chemotherapy for their metastatic pancreatic adenocarcinoma.
* Radical pancreatic resections (e.g. Whipple procedure) are not allowed < 6 months prior to randomization. Exploratory laparotomy, palliative (e.g. bypass) surgery, or other procedures (e.g. stents) are not allowed < 14 days prior to randomization. In any of the above cases, patients must be adequately recovered and stable prior to randomization.
* Prior treatment with > 6 cycles of traditional alkylating agent-based chemotherapy, > 2 cycles of carboplatin-based chemotherapy, prior treatment with irinotecan or oxaliplatin chemotherapy, or concurrent treatment with other experimental drugs or anti-cancer therapy.
* Curative radiation treatment to the pelvis or radiation therapy to ≥ 25% of bone marrow stores.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, short gut syndrome, or history of bowel obstruction due to peritoneal metastases.
* Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or non-melanoma skin cancer, unless at least 5 years have elapsed since last treatment and the patient is considered cured.
* Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, cerebrovascular diseases, uncontrolled hypertension, uncontrolled diabetes, uncontrolled psychiatric disorder, serious infection, active peptic ulcer disease, or other medical condition that may be aggravated by treatment.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Pre-existing neuropathy ≥ grade 2 from any cause.
* Patients with unstable metastasis to the central nervous system are excluded. Patients who have treated brain metastasis and are off steroids, anticonvulsants, and have documented stability of lesions for at least 3 months may be eligible. A CT scan or MRI is NOT required to rule out brain metastases unless there is clinical suspicion of CNS involvement.
* Pregnant or lactating women; women of child bearing potential must have a negative serum pregnancy test within 7 days of trial registration. Women or men of child bearing potential must use effective contraception (defined by the treating physician) which must be documented in study CRFs.
* Any other reason the investigator considers the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The difference Progression Free Survival (PFS) between Gemcitabine and FOLFOX treated patients in hENT1 high and hENT1 low pancreatic adenocarcinoma. | 2 Years
  Progression free survival will be measured from the date of diagnosis to the date of progression or death, patients who did not progress or is alive at the last date of follow-up will be censored for the analysis. Kaplan-Meier method will be used to estimate the survival function and log-rank test will be utilized to compare the study arms. The median PFS and the corresponding 95% confidence interval will be used for reporting purpose. The hazard ratio and the corresponding 95% two-sided confidence interval using Cox-proportional hazard regression will be presented.

SECONDARY OUTCOMES:
The difference in overall response rate (ORR) between the two treatment arms. | 2 years
The rate of disease control (DCR), defined as the sum of complete response rate (RR), partial RR, and stable disease between the two treatment arms. | 2 Years
The difference in overall survival (OS) between the two treatment arms. | 2 Years
Health-related quality of life (HRQL) parameters in patients with metastatic pancreas adenocarcinoma treated in both treatment arms. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Neil S. Chua, MD, FRCPC, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada